CLINICAL TRIAL: NCT01726075
Title: Neurodegeneration as Early Event in Pathogenesis of Diabetic Retinopathy:Multicentric, Prospective, Ph. II-III,Random.Controlled Trial to Assess Efficacy of Neuroprotective Drugs Administered Topically to Prevent/Arrest Diabetic Retinopathy
Brief Title: Trial to Assess the Efficacy of Neuroprotective Drugs Administered Topically to Prevent or Arrest Diabetic Retinopathy
Acronym: EUROCONDOR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: BCN Peptides (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4C-2011-02; 2012-001200-38 (EudraCT Number)
Record Dates: First submitted 2012-11-07; First posted 2012-11-14 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Diabetic Retinopathy
Keywords: diabetic retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- COLIRIOBCN070660 (Experimental): COLIRIOBCN070660 Somatostatin 1mg/mL Eye drops, solution. One drop/eye administered twice a day.
  Interventions: Drug: COLIRIOBCN070660
- Placebo (Placebo Comparator): Placebo Eye drops, solution. One drop/eye administered twice a day.
  Interventions: Drug: Placebo
- Brimonidine (Experimental): Brimonidine tartrate 2mg/mL One drop/eye administered twice a day.
  Interventions: Drug: Brimonidine

INTERVENTIONS:
Drug: COLIRIOBCN070660 — One drop per eye twice a day during 24 months
  Other Names: Somatostatin eye drops
  Arms: COLIRIOBCN070660
Drug: Placebo — One drop per eye twice a day during 24 months
  Other Names: placebo eye drops
  Arms: Placebo
Drug: Brimonidine — One drop per eye twice a day during 24 months
  Other Names: Brimonidine eye drops
  Arms: Brimonidine

SUMMARY:
To assess whether neuroprotective drugs administered topically (somatostatin and brimonidine) are able to prevent or arrest the development and progression of neurodegenerative changes

DETAILED DESCRIPTION:
To assess whether neuroprotective drugs administered topically (somatostatin and brimonidine) are able to prevent or arrest the development and progression of neurodegenerative changes related to diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type 2 diabetes mellitus
2. Diabetes duration ≥ 5 years
3. Aged between 45-75 years-old
4. ETDRS level < 20 (microaneurysms absent) (50% of enrolled patients) Or ETDRS levels 20 or 35 with presence of at least one microaneurysm in Field 2 between the superior and inferior arcades (50% of enrolled patients) in the Study Eye as determined by the Reading Centre.
5. Informed Consent

Exclusion Criteria:

1. Previous laser photocoagulation
2. Other diseases which may induce retinal degeneration (e.g. glaucoma)
3. Subject with a refractive error ≥ ± 5 diopter
4. Inadequate ocular media and/ or pupil dilatation that do not permit good quality fundus photography.
5. Renal failure (creatinine > 1.4 mg/dl)
6. HbA1C > 10 % in the previous 6 months and at Screening
7. Subjects taking somatostatin or brimonidine, for any indication, in the previous 3 months
8. Subject has a condition or is in a situation which may put the subject at significant risk, may confound the study results or may interfere significantly with the patient's participation in the study.
9. Pregnancy or nursing
10. Hypersensitivity to the active substances to be tested or to any of the excipients
11. Subject receiving systemic monoamine oxidase (MAO) inhibitor therapy or antidepressants which affect noradrenergic transmission (e.g. tricyclic antidepressants and mianserin)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2013-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Changes in the Implicit Time assessed by mfERG (IT-mfERG) at month 6, 12, 18 and 24 | month 24

SECONDARY OUTCOMES:
Retinal Nerve Fiber Layer (RNFL) assessed by Spectral Domain Optical Coherence Tomography (SD-OCT) at month 0 | month 0
Retinal Nerve Fiber Layer (RNFL) assessed by SD-OCT at month 6 | month 6
Retinal Nerve Fiber Layer (RNFL) assessed by SD-OCT at month 12 | month 12
Retinal Nerve Fiber Layer (RNFL) assessed by SD-OCT at month 18 | month 18
Retinal Nerve Fiber Layer (RNFL) assessed by SD-OCT at month 24 | month 24
Ganglion Cell Layer (GCL) assessed by SD-OCT at month 0 | month 0
Ganglion Cell Layer (GCL) assessed by SD-OCT at month 6 | month 6
Ganglion Cell Layer (GCL) assessed by SD-OCT at month 12 | month 12
Ganglion Cell Layer (GCL) assessed by SD-OCT at month 18 | month 18
Ganglion Cell Layer (GCL) assessed by SD-OCT at month 24 | month 24
Microaneurysm turnover assessed by Colour Fundus Photography (CFP - 45º/50º Field 2) at baseline | baseline
Microaneurysm turnover assessed by Colour Fundus Photography (CFP - 45º/50º Field 2) at month 6 | month 6
Microaneurysm turnover assessed by Colour Fundus Photography (CFP - 45º/50º Field 2) at month 12 | month 12
Microaneurysm turnover assessed by Colour Fundus Photography (CFP - 45º/50º Field 2) at month 18 | month 18
Microaneurysm turnover assessed by Colour Fundus Photography (CFP - 45º/50º Field 2) at month 24 | month 24
Retinal thickness assessed by SD-OCT at month 0 | month 0
Retinal thickness assessed by SD-OCT at month 6 | month 6
Retinal thickness assessed by SD-OCT at month 12 | month 12
Retinal thickness assessed by SD-OCT at month 18 | month 18
Retinal thickness assessed by SD-OCT at month 24 | month 24
Central retinal thickness assessed by SD-OCT at month 0 | month 0
Central retinal thickness assessed by SD-OCT at month 6 | month 6
Central retinal thickness assessed by SD-OCT at month 12 | month 12
Central retinal thickness assessed by SD-OCT at month 18 | month 18
Central retinal thickness assessed by SD-OCT at month 24 | month 24
Diabetic Retinopathy (DR) severity assessed by Early Treatment Diabetic Retinopathy Study (ETDRS) scale CFP - 30º/35º-7 fields at baseline | baseline
DR severity assessed by ETDRS scale CFP - 30º/35º-7 fields at month 24 | month 24

OTHER OUTCOMES:
Best Corrected Visual Acuity (BCVA) assessed by ETDRS scale at month 0 | month 0
BCVA assessed by ETDRS scale at month 6 | month 6
BCVA assessed by ETDRS scale at month 12 | month 12
BCVA assessed by ETDRS scale at month 18 | month 18
BCVA assessed by ETDRS scale at month 24 | month 24
Visual Fields defects assessed by Visual Fields Test at month 0 | month 0
Visual Fields defects assessed by Visual Fields Test at month 24 | month 24
Visual health assessed by Visual Function Questionnaire (VFQ-25) at month 0 | month 0
Visual health assessed by Visual Function Questionnaire (VFQ-25) at month 24 | month 24
Adverse Events assessed by inquiry at month 0 | month 0
Adverse Events assessed by inquiry at month 3 | month 3
Adverse Events assessed by inquiry at month 6 | month 6
Adverse Events assessed by inquiry at month 12 | month 12
Adverse Events assessed by inquiry at month 18 | month 18
Adverse Events assessed by inquiry at month 24 | month 24
ophthalmological examination: Refractive Error, Slit Lamp Exam, Ophthalmoscopy (Vitreous, Retina, Macula, Choroid, Optic Nerve), Intra-Ocular Pressure (IOP) Measurement at month 0 | month 0
ophthalmological examination: Refractive Error, Slit Lamp Exam, Ophthalmoscopy (Vitreous, Retina, Macula, Choroid, Optic Nerve), Intra-Ocular Pressure (IOP) Measurement at month 3 | month 3
ophthalmological examination: Refractive Error, Slit Lamp Exam, Ophthalmoscopy (Vitreous, Retina, Macula, Choroid, Optic Nerve), Intra-Ocular Pressure (IOP) Measurement at month 6 | month 6
ophthalmological examination: Refractive Error, Slit Lamp Exam, Ophthalmoscopy (Vitreous, Retina, Macula, Choroid, Optic Nerve), Intra-Ocular Pressure (IOP) Measurement at month 12 | month 12
ophthalmological examination: Refractive Error, Slit Lamp Exam, Ophthalmoscopy (Vitreous, Retina, Macula, Choroid, Optic Nerve), Intra-Ocular Pressure (IOP) Measurement at month 18 | month 18
ophthalmological examination: Refractive Error, Slit Lamp Exam, Ophthalmoscopy (Vitreous, Retina, Macula, Choroid, Optic Nerve), Intra-Ocular Pressure (IOP) Measurement at month 24 | month 24

CONTACTS AND LOCATIONS:
Overall Officials: José Cunha-Vaz, Prof., Principal Investigator — Association for Innovation and Biomedical Research on Light and Image
Locations (11):
- Syddansk Universitet (SDU), Odense, Denmark
- AP - Hopitaux de Paris (AP-HP), Paris, Paris, France
- Universitaet Ulm (UUlm), Ulm, Germany
- Italy (2):
  - Universita Vita-Salute San Raffaele (USR), Milan
  - Universita degli Study di Padova(UPadova), Padua
- Aibili - Cec, Coimbra, Coimbra District, Portugal
- Institut Catala de la Salut - Hospital Universitari Vall d'Hebron (ICS-HUVH), Barcelona, Barcelona, Spain
- United Kingdom (4):
  - Gloucestershire Hospitals NHS Foundation Trust (CHGH), Cheltenham, Gloucestershire
  - Moorfields Eye Hospital NHS Foundation Trust (MEH), London, London
  - Aston University (UAston)Heart of England NHS Foundation Trust, Birmingham
  - The University of Liverpool (UOL), Liverpool

REFERENCES:
- [Derived] Cunha-Vaz J, Ribeiro L, Costa M, Simo R. Diabetic Retinopathy Phenotypes of Progression to Macular Edema: Pooled Analysis From Independent Longitudinal Studies of up to 2 Years' Duration. Invest Ophthalmol Vis Sci. 2017 May 1;58(6):BIO206-BIO210. doi: 10.1167/iovs.17-21780. PMID 28785768
- [Derived] Santos AR, Ribeiro L, Bandello F, Lattanzio R, Egan C, Frydkjaer-Olsen U, Garcia-Arumi J, Gibson J, Grauslund J, Harding SP, Lang GE, Massin P, Midena E, Scanlon P, Aldington SJ, Simao S, Schwartz C, Ponsati B, Porta M, Costa MA, Hernandez C, Cunha-Vaz J, Simo R; European Consortium for the Early Treatment of Diabetic Retinopathy (EUROCONDOR). Functional and Structural Findings of Neurodegeneration in Early Stages of Diabetic Retinopathy: Cross-sectional Analyses of Baseline Data of the EUROCONDOR Project. Diabetes. 2017 Sep;66(9):2503-2510. doi: 10.2337/db16-1453. Epub 2017 Jun 29. PMID 28663190